CLINICAL TRIAL: NCT01354886
Title: A Phase I, Monocenter, Randomized, Placebo and Comparator Controlled, Single Blind, Rising Dose, Clinical Study to Determine Single Dose Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Four Doses of FSH-GEX™ According to Adaptive Design (25, 75, 150 and 300 IU) Administered Subcutaneously in Healthy Pituitary-suppressed Female Volunteers
Brief Title: Single Dose FSH-GEX™ in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glycotope GmbH (Industry)
Collaborators: Glycotope Biotechnology GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GEXGP240101
Record Dates: First submitted 2011-05-11; First posted 2011-05-17 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Female Infertility
Keywords: in-vitro fertilization; reproductive disorder
MeSH Terms: conditions — Infertility, Female | interventions — follitropin alfa; Urofollitropin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (7):
- FSH-GEX 25 IU (Experimental): 25 IU single dose
  Interventions: Drug: FSH-GEX™
- FSH-GEX 75 IU (Experimental): 75 IU single dose
  Interventions: Drug: FSH-GEX™
- FSH-GEX 150 IU (Experimental): 150 IU single dose
  Interventions: Drug: FSH-GEX™
- FSH-GEX 300 IU (Experimental): 300 IU single dose
  Interventions: Drug: FSH-GEX™
- Gonal-f (Active Comparator): 150 IU single dose
  Interventions: Drug: Gonal-f
- Bravelle (Active Comparator): 150 IU single dose
  Interventions: Drug: Bravelle
- Placebo (Placebo Comparator): single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FSH-GEX™ — single dose
  Other Names: follitropin epsilon
  Arms: FSH-GEX 150 IU; FSH-GEX 25 IU; FSH-GEX 300 IU; FSH-GEX 75 IU
Drug: Gonal-f — 150 IU single dose
  Other Names: follitropin alfa
  Arms: Gonal-f
Drug: Bravelle — 150 IU single dose
  Other Names: urinary FSH
  Arms: Bravelle
Drug: Placebo — single dose
  Arms: Placebo

SUMMARY:
The aim of the current study was the pharmacokinetic and pharmacodynamic characterization of a single dose administration of four doses of FSH-GEX™ in healthy pituitary-suppressed female volunteers, in comparison with two marketed comparator products.

DETAILED DESCRIPTION:
Healthy pituitary-suppressed female subjects received FSH-GEX™ (25, 75, 150 and 300 IU) in three of four possible ascending doses or one dose of two comparators (Bravelle® and Gonal-f®) and placebo in random order. The study consisted of three separate treatment periods. During each treatment period the subject received one single dose via a subcutaneous injection in the lower abdominal wall.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects from 18-40 years of age.
2. Subjects must be in good health.
3. Subjects must be willing to use additional non-hormonal contraception
4. Subjects must have used a combined oral contraceptive (COC) for at least one cycle.
5. Vital signs which are within the following ranges at baseline measurements: systolic blood pressure of 90-140 mmHg, diastolic blood pressure of 50-90 mmHg and pulse rate of 40 - 100 bpm.
6. Subjects must have a body weight of minimally 50.0 kg with a BMI between 18.0 and 29.0 kg/m^2 at baseline measurements.
7. Able to provide written informed consent prior to study participation.
8. Able to communicate well with the investigator and to understand and comply with the requirements of the study.

Exclusion Criteria:

1. Smokers of more than 10 cigarettes per day.
2. Average daily intake of more than 3 units of alcohol per day or an average weekly intake of more than 21 units alcohol.
3. Use of any prescription drug or ove the counter medication from screening until the end-of-study visit, without prior approval of the investigator.
4. Any drugs thay may reduce the effectiveness of COC from screening until the end-of-study visit.
5. Any follicle-stimulating hormone (FSH) preparation within 90 days prior to screening.
6. Administration of any investigational product or use of any investigational device within 30 days prior to screening.
7. Donation or loss of 500 mL or more blood within 90 days prior to first FSH-GEX™ dosing.
8. History of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated).
9. History of allergies for drugs, seafood, nuts, eggs, wasp-stings; history of atopic allergy (asthma, urticaria, eczematous dermatitis). A known hypersensitivity to any of the study drugs.
10. Any surgical or medical condition which might alter the absorption, distribution, metabolism, or excretion of drugs or which may jeopardize the subject in case of participation in the study.
11. History or presence of any malignancy.
12. Determined or suspected pregnancy.
13. Breast feeding women.
14. History of (or current) endocrine abnormalities.
15. Contraindication for the use of oral contraceptives.
16. Contraindication for the use of follitropin alfa, FSH or any of the excipients (hypersensitivity to follitropin alfa, FSH or any of the excipients; tumors of the hypothalamus or the pituitary gland; ovarian enlargement or cyst not due to polycystic ovarian disease; gynecological bleeding of unknown origin; ovarian, uterine, or mammary carcinoma).
17. Porphyria or family history of porphyria.
18. History of ovarian surgery.
19. Any ovarian or abdominal abnormality that would interfere with adequate ultrasound investigation.
20. An abnormal cervical smear.
21. History or presence of an immune-compromising disease, or a positive human immunodeficiency virus (HIV) test result in the past or at the screening visit.
22. History of Hepatitis B or C, or a positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result at the screening visit.
23. History of drug or alcohol abuse within the 12 months prior to the screening visit or evidence of such abuse.
24. Planned surgery or hospitalization during the period of the study.
25. Concurrent participation or participation within 30 days before screening in another clinical trial, or participation in more than 3 clinical studies within 12 months, prior to the expected date of enrolment into the study.
26. Injection of one or more doses of any depot contraceptive drug /drug combination or hormonal implants <= 10 months prior to screening.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
to assess the safety and (local) tolerability of FSH-GEX™ following single rising dose administration by subcutaneous injection | up to 87 days
  frequency of dose related adverse events, measurement of vital signs, body measurements, transvaginal ultrasound, ECG and laboratory values in comparison to placebo and the two comparators with marketing authorization
to determine FSH pharmacokinetic parameters of FSH-GEX™ following single dose administration by subcutaneous injection (part 1) | before FSH/Placebo administration until 240 hours thereafter
  Peak plasma concentration (Cmax)
to determine FSH pharmacokinetic parameters of FSH-GEX™ following single dose administration by subcutaneous injection (part 2) | before FSH/Placebo administration until 240 hours thereafter
  Area under the plasma concentration versus time curve (AUC)

SECONDARY OUTCOMES:
to assess the pharmacodynamic effect of FSH-GEX™ following single rising dose administration by subcutaneous injection (part 1) | before FSH/Placebo administration until 240 hours thereafter
  determined by Estradiol (E2) and inhibin B concentrations depending on dose
to assess the pharmacodynamic effect of FSH-GEX™ following single rising dose administration by subcutaneous injection (part 2) | up to a maximum of 87 days
  ovarian follicle number and size as determined by transvaginal ultrasonography depending on dose

CONTACTS AND LOCATIONS:
Overall Officials: Glycotope GmbH, Study Director — Glycotope GmbH
Locations (1):
- Glycotope Investigational Site, Groningen, Netherlands

REFERENCES:
- [Result] Abd-Elaziz K, Duijkers I, Stockl L, Dietrich B, Klipping C, Eckert K, Goletz S. A new fully human recombinant FSH (follitropin epsilon): two phase I randomized placebo and comparator-controlled pharmacokinetic and pharmacodynamic trials. Hum Reprod. 2017 Aug 1;32(8):1639-1647. doi: 10.1093/humrep/dex220. PMID 28591833